Official Title: A MULTIPLE-CENTER, MULTIPLE-DOSE AND REGIMEN,

RANDOMIZED, ACTIVE COMPARATOR CONTROLLED, DOUBLE-

MASKED, PARALLEL GROUP, 36 WEEK STUDY TO

INVESTIGATE THE SAFETY, TOLERABILITY,

PHARMACOKINETICS, AND EFFICACY OF RO6867461 ADMINISTERED INTRAVITREALLY IN PATIENTS WITH

CHOROIDAL NEOVASCULARIZATION SECONDARY TO AGE-

RELATED MACULAR DEGENERATION

NCT Number: NCT02484690

**Document: STATISTICAL ANALYSIS PLAN** 

Version & Date: Version 1: 13-Feb-2017

## STATISTICAL ANALYSIS PLAN SIGNATURE PAGE

Upon review of this document, the undersigned approves this version of the Statistical Analysis Plan, authorizing that the content is acceptable for the reporting of this study.

## Statistical Analysis Plan V1.0 for Protocol BP29647.

| | Name | Signature | Date |
|--------------|-----------------------|-----------|-----------|
| Author: | | | 14FEB2017 |
| Position: | Statistical Scientist | | |
| Company: | F. Hoffmann-La Roche | e Ltd. | |
| | Name | Signature | Date |
| Approved By: | | | FEB2017 |
| Position: | | | |
| Company: | F. Hoffmann-La Roche | e Ltd. | |

## STATISTICAL ANALYSIS PLAN

TITLE:

A MULTIPLE-CENTER, MULTIPLE-DOSE AND

REGIMEN, RANDOMIZED, ACTIVE COMPARATOR

CONTROLLED, DOUBLE-MASKED, PARALLEL GROUP,

36 WEEK STUDY TO INVESTIGATE THE SAFETY,

TOLERABILITY, PHARMACOKINETICS, AND EFFICACY OF RO6867461 ADMINISTERED INTRAVITREALLY IN PATIENTS WITH CHOROIDAL NEOVASCULARIZATION

**SECONDARY TO AGERELATED MACULAR** 

DEGENERATION

PROTOCOL NUMBER:

BP29647

STUDY DRUG:

RO687461

**VERSION NUMBER:** 

1.0

IND NUMBER:

119225

**EUDRACT NUMBER:** 

N/A

SPONSOR:

F. Hoffmann-La Roche Ltd

**PLAN PREPARED BY:** 

**DATE FINAL:** 

13 February 2017

## STATISTICAL ANALYSIS PLAN SIGNATURE PAGE

Upon review of this document, the undersigned approves this version of the Statistical Analysis Plan, authorizing that the content is acceptable for the reporting of this study.

## Statistical Analysis Plan V1.0 for Protocol BP29647.

| | Name | Signature | Date |
|-----------|-----------------------|-----------|-----------|
| Author: | | | 14FEB2017 |
| Position: | Statistical Scientist | | |
| Company: | F. Hoffmann-La Roc | he Ltd. | |

| | Name | Signature | Date |
|-----------------|--------------------|-----------|------------|
| Approved<br>By: | | | 14 FEB2017 |
| Position: | | | |
| Company: | F. Hoffmann-La Roc | he Ltd. | |

## **TABLE OF CONTENTS**

| | Statistical An | alysis Plan Signature Page | 2 |
|---|---|---|---|
| 1. | BACKGROU | ND | 5 |
| 2. | STUDY DES | IGN | 5 |
| | 2.1 | Protocol Synopsis | е |
| | 2.2 | Outcome Measures | 6 |
| | 2.2.1 | Primary Efficacy Outcome Measures | 6 |
| | 2.2.2 | Secondary Efficacy Outcome Measures | 6 |
| | 2.2.3 | Exploratory Efficacy Outcome Measures | 6 |
| | 2.2.4 | Pharmacokinetic Efficacy Outcome Measures | 8 |
| | 2.2.5<br>Measures | Pharmacodynamic Biomarker Outcome<br>8 | |
| | 2.2.6 | Safety Outcome Measures | 8 |
| | 2.3 | Determination of Sample Size | 8 |
| | 2.3.1<br>Population | Sample Size and Power for Treatment-Naive Evaluation | 8 |
| | 2.3.2<br>Incomplete | Sample Size and Power for anti-VEGFResponder Population Evaluation | g |
| | 2.4 | Analysis Timing | 9 |
| 3. | STUDY CON | IDUCT | g |
| | 3.1 | Randomization | 9 |
| | 3.2 | Internal Review Committee | 10 |
| | 3.3 | Data Monitoring | 10 |
| 4. | STATISTICA | IL METHODS | 10 |
| | 4.1 | Analysis Populations | 10 |
| | | Efficacy, Pharmacokinetic, and dynamic Population | 10 |
| | | Population A: All Patient Randomized to Arms, and D | 10 |
| | 4.1.1.2<br>A and E | Population B: All Patients Randomized to Arms 10 | |
| | Populat | Population C: Anti-VEGF-Incomplete Responder tion | 11 |
| | 867461—F. Hof | fmann-La Roche Ltd<br>Ian BP29647 | |

| 4.1.2 | Safety Population11 |
|---|---|
| 4.2 | Analysis of Study Conduct11 |
| 4.3 | Analysis of Treatment Group Comparability11 |
| 4.4 | General Considerations11 |
| 4.4.1 | Visit Windows11 |
| 4.4.2 | Baseline12 |
| 4.5 | Efficacy Analysis12 |
| 4.5.1 | Primary Efficacy Endpoint12 |
| 4.5.1.1 | Evaluation in the Treatment-Naive Population12 |
| 4.5.1.2<br>Respon | Evaluation in the anti-VEGF Incomplete der Population C13 |
| 4.5.2 | Secondary Efficacy Endpoints13 |
| 4.5.3 | Exploratory Efficacy Endpoints14 |
| 4.5.4 | Sensitivity Analyses14 |
| 4.5.5 | Subgroup Analyses14 |
| 4.6 | Safety Analyses15 |
| 4.6.1 | Adverse Events15 |
| 4.6.2 | Clinical Laboratory Test Results15 |
| 4.6.2.1<br>Transfo | Standard Reference Ranges and brmation of Data15 |
| 4.6.2.2 | Definition of Laboratory Abnormalities16 |
| 4.6.3 | Vital Signs16 |
| 4.6.4 | ECG Data Analysis16 |
| 4.6.5 | Anti-Drug Antibody Data Analysis16 |
| 4.6.6 | Ocular Assessments16 |
| 4.6.7 | Concomitant Medications17 |
| 4.6.8 | Exposure to Study Medication17 |
| 4.7 | Missing Data17 |
| 4.8 | Interim Analyses17 |
| | LIST OF TABLES |
| Figure 1 Stu | udy Design5 |
| RO6867461—F. Hof<br>Statistical Analysis P | fmann-La Roche Ltd<br>Ian BP29647 |

## 1. <u>BACKGROUND</u>

This Statistical Analysis Plan (SAP) documents the statistical methods for summarizing and analyzing the efficacy and safety data from study BP29647. The main purpose of this SAP is to describe the data handling rules, derivation rules, and statistical analysis methods.

## 2. STUDY DESIGN

This is a multiple-center, multiple-dose and regimen, randomized, active comparator controlled, double-masked, five parallel groups, 36-week study in patients with subfoveal CNV secondary to AMD. The study design is shown in Figure 1 Study Design.

The five groups of this study are as follows.

- Arm A: 0.5 mg ranibizumab IVT every 4 weeks for 32 weeks (9 injections)
- Arm B: 1.5 mg RO6867461 IVT every 4 weeks for 32 weeks (9 injections)
- Arm C: 6 mg RO6867461 IVT every 4 weeks for 32 weeks (9 injections)
- Arm D: 6 mg RO6867461 IVT every 4 weeks up to Week 12 (4 injections), followed by 6 mg RO6867461 IVT every 8 weeks (i.e., on Weeks 20 and 28; 2 injections)
- Arm E: 0.5 mg ranibizumab IVT every 4 weeks up to Week 8 (3 injections), followed by 6 mg RO6867461 IVT every 4 weeks (6 injections)



Figure 1 Study Design

Q4W = every 4 weeks; Q8W = every 8 weeks

These treatment arms have been chosen to compare the treatments in a treatment-naïve population and in an anti-VEGF-incomplete-responder population. For the treatment-naïve population the arms B and C will be compared with the reference arm A. For the anti-VEGF incomplete responder population, a subgroup of arm E will be compared to a similar subgroup of arm A.

#### 2.1 PROTOCOL SYNOPSIS

The Protocol Synopsis is in Appendix 1. For additional details, see the Schedule of Assessments in Appendix 2.

#### 2.2 OUTCOME MEASURES

For efficacy analyses only measurements in the study eye are used; except where explicitly stated.

For safety analyses events and measurements in both eyes will be included in the analyses, except for imaging.

## 2.2.1 Primary Efficacy Outcome Measures

The primary efficacy outcome measure is the mean change from baseline in BCVA at Week 36 using the ETDRS modified charts.

## 2.2.2 <u>Secondary Efficacy Outcome Measures</u>

The secondary efficacy outcome measures include functional (BCVA) and anatomical PD imaging measures relevant to the mechanism of action of RO6867461 as follows.

#### BCVA:

- Proportion of patients gaining ≥15 letters from baseline in BCVA at Week 36
- Proportion of patients with BCVA of 20/40 or better at Week 36
- Proportion of patients with BCVA of 20/200 or worse at Week 36

Anatomic outcome measures by SD-OCT:

- Mean change from baseline in foveal center point thickness at Week 36
- Mean change from baseline in mean CST (1 mm diameter) at Week 36
- Proportion of patients with no intraretinal fluid, subretinal fluid, cysts, or pigment epithelial detachment at Week 36 (dry retina definition No1)

Anatomic outcome measures by FFA:

- Mean change from baseline in total area of CNV at Week 36
- Mean change from baseline in total area of CNV component at Week 36
- Mean change from baseline in total area of leakage at Week 36

## 2.2.3 <u>Exploratory Efficacy Outcome Measures</u>

The exploratory outcome measures for this study are the following:

- Proportion of patients gaining 5 or more, 10 or more, and 30 or more letters in BCVA on ETDRS charts over time
- Proportion of patients losing 5 or more, 10 or more, 15 or more, and 30 or more letters in BCVA on ETDRS charts over time

· Proportion of patients with resolution of RAP and PCV (ICGA) over time

Combined dry retina outcome measures:

- Proportion of patients with absence of IRF, SRF and cysts all by SD-OCT, and leakage by FFA at Weeks 12, 24 and 36 (dry retina definition No2)
- Proportion of patients with absence of IRF, SRF, cysts and PED all by SD-OCT at Weeks 12, 24 and 36 (dry retina definition No3)

Individual dry retina outcome measures:

- Proportion of patients with absence of IRF (by SD-OCT) over time
- · Proportion of patients with absence of SRF (by SD-OCT) over time
- · Proportion of patients with absence of cysts (by SD-OCT) over time
- · Proportion of patients with absence of PED (by SD-OCT) over time
- Proportion of patients with absence of leakage (by FFA) over time

Table 1 Description of Secondary Outcome Measures

| Secondary<br>Endpoint | Detailed Definition | Variable names used by central reading center (and combinations therefore for certain endpoints) |
|---|---|---|
| foveal center point<br>thickness | Thickness from Inner Limiting Membrane to the Retinal Pigment Epithelial at the horizontal slice closest to the center of the fovea | OCTcentralretinalthickness (SDTM variables : CENT RET THICK R1-3) |
| mean CST | Mean thickness from Inner<br>Limiting Membrane to the Retinal<br>Pigment Epithelial over the 1 mm<br>central subfield | OCTCentralSubfieldThickness (SDTM variables: CENT SUBFIELD THICK ILM-RPE R1-3) |
| intra-retinal fluid<br>(IRF) | Presence of fluid within the retina | OCTIntraRetinalFluid (SDTM variable: INTRARETINAL FLUID) |
| cysts | Presence of cystoid space (fluid) in the retina | OCTCystoidSpaces (SDTM variable:<br>CYSTOID SPACES) |
| sub-retinal fluid<br>SRF) | Presence of fluid between the retina and the retinal pigment epithelium | OCTSubretinalFluidThicknessNotPresent<br>(derived from SDTM variable: Subret Fluid<br>Thick) |
| pigment epithelial<br>detachment (PED) | Presence of a detachment of the pigment epithelium from the Bruch's membrane Dry retina Definition 1: | OCTPigmentEpithelialDefectThickness (SDTM variables: PED THICK R1-3) |
| area of CNV | Total area of CNV lesion | FATotalLesionSizeMM (SDTM variables; FA TOTAL LESION SIZE R1-3) |
| area of CNV component | Total area of CVN membrane | FAArea (SDTM variable: FA CNV SIZE R1-3) |
| total area of | Total area of fluorescein | FALeakage (SDTM variable: FA |

| leakage | leakage | LEAKAGE R1-3) |
|---------|---------|---------------|

- Biomarkers in plasma related to angiogenesis and inflammation: Ang-1, Tie-2, VEGFR, PLGF, bFGF, PDGF, IL-1b, IL-6, eotaxin, autotaxin
- Pro-angiogenic factors in aqueous humor and vitreous samples for patients who
  provide additional consent to participate.

## 2.2.4 Pharmacokinetic Efficacy Outcome Measures

The pharmacokinetic (PK) outcome measures for this study are as follows:

 PK profiles and parameters derived from the nonlinear mixed effects modeling approach following IVT administration of RO6867461, including the following parameters:

Primary parameters: CL and V

Secondary parameters: C<sub>max</sub>, AUC<sub>inf</sub>, AUC<sub>0-t</sub>, t<sub>max</sub>, t<sub>1/2</sub>

Compartmental analysis to assess IVT concentrations, as appropriate (exploratory)

RO6867461 concentrations in aqueous humor samples for patients who provide additional consent to participate (exploratory)

## 2.2.5 Pharmacodynamic Biomarker Outcome Measures

Plasma biomarker outcome measures for this study are as follows:

Change in plasma levels of VEGF and Ang-2

## 2.2.6 Safety Outcome Measures

The safety outcome measures for this study are as follows:

- Incidence and severity of ocular adverse events
- Incidence and severity of non-ocular adverse events
- Incidence of laboratory abnormalities, based on hematology, clinical chemistry, and urinalysis test results
- Incidence of anti-RO6867461 antibodies
- ECGs
- Vital signs
- · Other safety biomarkers

## 2.3 DETERMINATION OF SAMPLE SIZE

# 2.3.1 <u>Sample Size and Power for Treatment-Naive Population Evaluation</u>

The sample size for the treatment-naive population is based on the primary efficacy outcome of mean change in BCVA from baseline to Week 36. Each RO6867461 dose or dose regimen group (Arms B, C, and D) will be compared to the control group (Arm A).

Consider 68 patients randomized to Arm A and 45 randomized to each of Arms B, C, and D, with a drop-out rate of 10%. Assuming a standard deviation of 13.5 letters, this sample size would provide approximately 80% power to detect a true difference of 5.9 letters at the one-sided  $\alpha$  level of 10%. The minimum detectable difference would be approximately 3.5 letters.

## 2.3.2 <u>Sample Size and Power for anti-VEGF-Incomplete-Responder</u> Population Evaluation

The sample size for anti-VEGF-incomplete-responder population is based on the primary efficacy outcome of mean change in BCVA from Week 12 to Week 36 in the subset of anti-VEGF-incomplete-responders, between Arm A and Arm E.

Consider 68 patients randomized to both Arms A and E with 65% meeting the criteria for inclusion in anti-VEGF–incomplete-responder subgroup and a drop-out rate of 10%. Assuming a standard deviation of 9.7 letters, this sample size would provide approximately 80% power to detect a true different of 4.7 letters at the one-sided  $\alpha$  level of 10%. The minimum detectable difference would be approximately 2.7 letters.

#### 2.4 ANALYSIS TIMING

The primary analysis will be performed at the end of the study, after the last patient has completed Week 36 final visit.

## 3. STUDY CONDUCT

## 3.1 RANDOMIZATION

After written informed consent has been obtained, all patients will receive a screening number assigned through the Interactive Voice and Web Response System (IxRS). After all patient eligibility requirements are confirmed on Day 1 visit the site personnel will contact the IxRS for assignment of a patient identification number (a separate number from the screening number).

Patients will be randomized in a 3:2:2:2:3 ratio to one of the study treatment arms A, B, C, D or E (see 2 for details):

Patients will be randomized on the same day the study treatment is to be initiated (Day 1 visit). After randomization and at each visit with study treatment administration (i.e., including Day 1) the IxRS will assign the appropriate study treatment kit to be used.

Randomization will be stratified for the two factors below:

- Baseline BCVA ETDRS letter score assessed on Day 1 (69 letters or better vs.
   68 letters or worse)
- Presence/absence of retinal angiomatous proliferation (RAP) or polypoidal choroidal vasculopathy (PCV) at screening as assessed by the Reading Center

## 3.2 INTERNAL REVIEW COMMITTEE

A Roche internal monitoring committee (IMC) will be responsible in the event of an interim analysis for sample size evaluation, operational/administrative purposes, and/or for safety data monitoring. For other objectives, the IMC will review the safety data and will be responsible for evaluating efficacy data for instance where assessment of benefit-risk is warranted. These analyses will take place at predefined time points or on an ad-hoc basis.

The IMC consists of a selected subset of Roche representatives including a biostatistician, safety representative, clinical science representative, clinical pharmacology representative, and pharmacometrician. The IMC members participating in a given interim analysis will be kept to the minimum required to address the objective of that interim analysis. Additional Roche Representatives might be involved to produce/process the unmasked listing/data to be analyzed by the IMC.

Full details regarding the IMC will be provided separately in the IMC agreement.

## 3.3 DATA MONITORING

An IMC will review safety data, and may review efficacy data to assess benefit-risk.

## 4. STATISTICAL METHODS

## 4.1 ANALYSIS POPULATIONS

The following analysis populations will be defined: "Efficacy, Pharmacokinetic, and Pharmacodynamic Population" and safety population.

## 4.1.1 <u>Efficacy, Pharmacokinetic, and Pharmacodynamic</u> Population

All randomized patients will be included in the efficacy, PK, and PD analysis population. Patients who receive study drug in the study eye different that to which they were randomized will be included in the group to which they were randomized.

## 4.1.1.1 Population A: All Patient Randomized to Arms A, B, C, and D

Population A consists of all patients randomized to the treatment arms A, B, C and D. In this population, the baseline reference is the latest non-missing observation before start of study treatment. Population A will be used for the evaluation of efficacy in the treatment-naive population.

## 4.1.1.2 Population B: All Patients Randomized to Arms A and E

Population B consists of all patients randomized to the treatment arms A and E. For this population, the Week 12 visit is the baseline for all efficacy and PD analyses. Therefore, the primary endpoint is BCVA change from Week 12. A subgroup of Population B, Population C, will be used for the evaluation of efficacy in the anti-VEGF-incomplete- responder population and is defined below.

## 4.1.1.3 Population C: Anti-VEGF-Incomplete Responder Population

The primary anti-VEGF-incomplete responder population is defined as subpopulation of population B consisting of

 Population C: Patients in population B with BCVA ≤ 68 at Week 12 with at least one letter improvement relative to baseline.

Additional exploratory anti-VEGF-incomplete responder populations are defined as

- Population C1: Patients in population B with improvement of less than 15 letters at Week 12
- Population C2: Patients in population B without dry retina at Week 12 (dry retina definition No 2)

## 4.1.2 Safety Population

All patients who have received at least one dose of the study treatment, whether prematurely withdrawn from the study or not, will be included in the safety analysis for this population. Patients who receive study drug in the study eye different from which they were randomized to will be included into the group to which their treatment profile match best.

#### 4.2 ANALYSIS OF STUDY CONDUCT

The number of patients who are enrolled, discontinued, and completed the study will be summarized as well as the major protocol violations. Demographic and baseline characteristics will be summarized with descriptive statistics. The analysis will be performed for populations A and C.

## 4.3 ANALYSIS OF TREATMENT GROUP COMPARABILITY

Demographics, baseline characteristics (including ocular assessments, patient disposition, and medical history), and all baseline laboratory values will be summarized descriptively by treatment arm using frequency tables and summary statistics providing means, medians, standard deviations, first and third quartiles, and extreme values.

## 4.4 GENERAL CONSIDERATIONS

## 4.4.1 Visit Windows

Visit windowing will be performed for this study with nominal visits/assessments falling outside of allowable protocol-defined visit windows, being reassigned to an appropriate visit for use in analyses.

If multiple valid (non-missing) values for a variable are recorded in the same visit window, one record will be selected for summary/analysis of the data by the following priority:

· The originally scheduled visit assessment

· The assessment closest to the target assessment day.

If scheduled assessments were grouped into multiple visits, the assessments will be assigned to a single visit provided all assessments fall within the same visit window.

Note that unscheduled visits could potentially be included in summaries and analyses following the application of these visit assignment rules.

Assessments that fall outside of the protocol-defined visit windows will be assigned to the closest target visit.

Unless otherwise specified, all analyses and summaries involving visit, will use visits assigned after visit windowing has been performed.

## 4.4.2 Baseline

For the evaluation in the treatment-naive population, the baseline measurement is the latest non-missing observation before the first dose of study medication. For the evaluation in the anti-VEGF-incomplete-responder population, the baseline is the observation from Study Week 12. If the week 12 observation is missing, the patient will not be included in the incomplete responder population. For patients who did not receive any study medication, baseline will be set as the last available assessment before and including day 1.

#### 4.5 EFFICACY ANALYSIS

The List of Planned Outputs (LoPO) contains the full list of reports for the efficacy analysis.

## 4.5.1 <u>Primary Efficacy Endpoint</u>

## 4.5.1.1 Evaluation in the Treatment-Naive Population

For the evaluation of efficacy in the treatment-naïve population, all patients in Population A will be used.

The primary efficacy variable is the BCVA change from baseline to Week 36. The primary efficacy analysis will be performed using a Mixed Model for Repeated Measurement (MMRM) model. The model will include the categorical covariates of randomization stratification indicator for presence of RAP or PCV, treatment group, visit, and visit by treatment group interaction and the continuous covariate of baseline BCVA. An unstructured variance-covariance model will be used to account for within-patient correlation, but another variance-covariance structure, such as AR(1), may be used in case of convergence issues.

In case of a significant departure from the normality assumptions required for the MMRM, a nonparametric Mann-Whitney  $\boldsymbol{U}$  test will be used to compare change from baseline between treatment arms at given visits.

The primary statistical tests will test the null hypotheses:

H<sub>0</sub>: no difference between each of the treatment group (Arms B, C, or D) and the control group (Arm A), in mean BCVA change from baseline to Week 36 vs.

H<sub>A</sub>: Arms B, C or D means are different from Arm A mean.

The model-based estimate of the difference between each of the treatment group (Arms B, C, and D) and the control group (Arm A) at Week 36, together with 95% confidence intervals and corresponding p-value will be reported as the primary efficacy measures in this population.

The mean and 95% confidence interval (CI) within each treatment group and for the difference in change from baseline between RO6867461 treatment groups (Arms B, C, and D) and the control group (Arm A) at the other time-points will also be reported. There will be no formal correction for multiple comparisons.

For the primary endpoints, a statistically significant difference at week 36 between any of the treatment Arms B, C, or D and Arm A will be concluded if the corresponding unadjusted 2-sided p-value is below 0.2.

## 4.5.1.2 Evaluation in the anti-VEGF Incomplete Responder Population C

For the evaluation of efficacy in the anti-VEGF-incomplete-responder all patients in the population C will be used.

The primary efficacy variable is BCVA change from Week 12 to Week 36. The primary efficacy analysis will be performed using a MMRM model described in section 4.5.1.1.

The model-based estimate of the difference in change from baseline between the treatment group (Arm E) and the control group (Arm A) means at Week 36, together with 95% Confidence and corresponding p-value will be reported as the primary efficacy measure in this population.

The mean and 95% confidence intervals within each treatment group and for the difference between RO6867461 treatment group and the control group change from baseline at the other time points will also be reported. There will be no formal correction for multiple comparisons.

## 4.5.2 <u>Secondary Efficacy Endpoints</u>

All analyses of secondary efficacy endpoints as defined in section 2.2.2 will be performed for population A and for population C, using their respective baseline definition (see 4.4.2).

For all secondary endpoints measured on a continuous scale, the same MMRM model used for the change from baseline BCVA will be employed. Nominal p-values for treatment effect will be reported for all post-baseline visits without correction for multiple testing.

Binary endpoints will be analyzed using Generalized Estimating Equations (GEE) with a binomial distribution, logit link function for odds ratios and identity link for risk differences, and unstructured covariance. In case of convergence issues, other covariance structures, such as AR(1) covariance structure, will be used.

The model will include the categorical covariates of treatment group, visit, and visit by treatment group interaction and randomization stratification indicator for presence of RAP or PCV and the continuous covariate of baseline outcome measure.

Least squares means on the probability scale for each treatment arm with the corresponding 95% confidence intervals and odds ratios relative to the control arm will be computed for all post-baseline visits.

Data transformation (e.g., logarithmic transformation) may be applied as appropriate. Other statistical models and additional analyses may also be performed as appropriate. Fisher's exact test may be used for binary endpoints in case GEE models do not converge.

In addition, the influence of baseline parameters will be evaluated as covariates in the MMRM model and in subgroup analysis as appropriate (see Section 4.5.5).

## 4.5.3 Exploratory Efficacy Endpoints

Additional exploratory analyses may be performed as warranted in order to more fully understand the relationship over time between parameters and either nominal dose or concentration of RO6867461. They will be described here.

- Proportion of patients with resolution of PCV over time
- · Proportion of patients with resolution of RAP over time

## 4.5.4 Sensitivity Analyses

Effects of prognostic factors on the BCVA change from baseline will be investigated using the MMRM model described in section 4.5.1. The measurement at BL (baseline) of each of the following variables may be used as covariates in the model:

- Age
- CNV component area, (FFAArea)
- LLD (Difference between BCVATOT for the BCVA assessment and LLVATOT for the LLVA assessment)

The sensitivity analyses will be performed separately for each covariate in populations A and C.

## 4.5.5 Subgroup Analyses

For the sub-group analysis the MMRM for change from baseline in BCVA will be used in the following subgroups:

Gender

- CNV lesion type at baseline (FACNV) CNV on FA as Classic, Classic+occult or Occult
- CNV lesion type by ICG at baseline as 3 categories: PCV, RAP or Neither
- OCT analysis: Fluid Type at baseline (by type of fluid intraretinal, subretinal or other)
- BCVA Categories at baseline (20/40 or better vs worse than 20/40, 20/200 or better vs worse than 20/200),
- · Baseline LLD quartiles or medians.

The subgroup analyses will be performed separately for each sub-group factor in populations A and C. For population C the subgroups will be defined based on the baseline defined for this population. Subgroup analyses in population C will be performed only if there are a sufficient number of patients in this population.

## 4.6 SAFETY ANALYSES

All safety analyses will be based on the safety analysis population. The LoPO contains the full list of reports for safety analyses.

## 4.6.1 Adverse Events

The original terms recorded on the eCRF by the Investigators for adverse events will be standardized by the Sponsor. Adverse events will be summarized by mapped term and appropriate thesaurus level, including a separate summaries for ATE events (see <u>Appendix 3</u>).

Separate summaries will be prepared for systemic and ocular adverse events, with events in the study eye and non-study eye summarized separately. SAEs will be summarized similarly. Adverse events leading to discontinuation from the study will be listed and tabulated.

## 4.6.2 <u>Clinical Laboratory Test Results</u>

All clinical laboratory data will be stored on the database in the units in which they were reported. Patient listings and summary statistics at each assessment time will be presented using the International System of Units (SI units; Système International d'Unités). Laboratory data not reported in SI units will be converted to SI units before processing.

Laboratory test values will be presented by individual listings with flagging of values outside the normal ranges.

## 4.6.2.1 Standard Reference Ranges and Transformation of Data

Roche standard reference ranges, rather than the reference ranges of the Investigator, will be used for all parameters. For most parameters, the measured laboratory test result will be assessed directly using the Roche standard reference

range. Certain laboratory parameters will be transformed to Roche's standard reference ranges.

A transformation will be performed on certain laboratory tests that lack sufficiently common procedures and have a wide range of Investigator ranges, e.g., enzyme tests that include AST, ALT, and alkaline phosphatase and total bilirubin. Given that the standard reference ranges for these parameters have a lower limit of zero, only the upper limits of the ranges will be used in transforming the data.

## 4.6.2.2 Definition of Laboratory Abnormalities

For all laboratory parameters included, there exists a Roche predefined standard reference range. Laboratory values falling outside this standard reference range will be labeled "H" for high or "L" for low in patient listings of laboratory data.

In addition to the standard reference range, a marked reference range has been predefined by Roche for each laboratory parameter. The marked reference range is broader than the standard reference range. Values falling outside the marked reference range that also represent a defined change from baseline will be considered marked laboratory abnormalities (i.e., potentially clinically relevant). If a baseline value is not available for a patient, the midpoint of the standard reference range will be used as the patient's baseline value for the purposes of determining marked laboratory abnormalities. Marked laboratory abnormalities will be labeled in the patient listings as "HH" for very high or "LL" for very low.

## 4.6.3 Vital Signs

Vital signs data will be presented by individual listings with flagging of values outside the normal ranges and flagging of marked abnormalities. In addition, tabular summaries will be used, as appropriate.

## 4.6.4 ECG Data Analysis

ECG data will be presented by individual listings with flagging of values outside the normal ranges and flagging of marked abnormalities. In addition, tabular summaries will be used, as appropriate.

## 4.6.5 Anti-Drug Antibody Data Analysis

The number and percentage of patients who test positive for plasma antibodies to RO6867461 at baseline and at the study visits will be tabulated, but not for treatment arm A.

## 4.6.6 Ocular Assessments

Results of the following ocular assessments will be summarized by time point for the study eye using descriptive summaries: BCVA (also for the non-study eye), IOP (also for the non-study eye), and changes from baseline in these measurements will be tabulated.

## 4.6.7 Concomitant Medications

The original terms recorded on the patients' eCRF by the Investigator for concomitant medications will be standardized by the Sponsor by assigning preferred terms.

Concomitant medications will be presented in summary tables and listings.

## 4.6.8 Exposure to Study Medication

The following extent to study medication will be summarized by treatment arm:

- Duration of treatment, to be calculated as first day to last day to masked study medication
- Relative extent of exposure as number of given intravitreal injections divided by number of planned intravitreal injections of masked study medication during the treatment duration of a patient.

## 4.7 MISSING DATA

An analysis of the sensitivity of the assumptions on missing values may be performed for the primary efficacy variable.

The primary endpoint analysis using the MMRM assumes a missing at random (MAR) missing-data mechanism (i.e., the probability that missing data are dependent on other observed variables, but not on the missing data itself.)

A LOCF imputation will be applied to the primary end-point as a sensitivity analysis.

## 4.8 INTERIM ANALYSES

Given the hypothesis-generating nature of this study, the Sponsor may conduct up to two additional interim analyses of efficacy. The decision to conduct such an interim analysis and its timing will be documented in the Sponsor's study master file prior to the conduct of the interim analysis. The Clinical Study Report will also document that such an interim analysis occurred. The interim analysis, should it occur, will be performed and interpreted by members of the IMC and DRC who would then be unmasked at the treatment group level. Access to treatment assignment information will follow the Sponsor's standard procedures.

Details of the interim analyses are described in the IMC charter.

## Appendix 1

## **SYNOPSIS OF PROTOCOL NUMBER BP29647**

| TITLE | A MULTIPLE-CENTER, MULTIPLE-DOSE AND REGIMEN, RANDOMIZED, ACTIVE COMPARATOR CONTROLLED, DOUBLE-MASKED, PARALLEL GROUP, 36-WEEK STUDY TO INVESTIGATE THE SAFETY, TOLERABILITY, PHARMACOKINETICS, AND EFFICACY OF RO6867461 ADMINISTERED INTRAVITREALLY IN PATIENTS WITH CHOROIDAL NEOVASCULARIZATION SECONDARY TO AGE-RELATED MACULAR DEGENERATION |
|---|---|
| PROTOCOL NUMBER: | BP29647 |
| VERSION: | 3 |
| EUDRACT NUMBER: | N/A |
| IND NUMBER: | 119225 |
| TEST PRODUCT: | RO6867461 |
| PHASE: | 11 |
| INDICATION: | Choroidal neovascularization (CNV) secondary to agerelated macular degeneration (AMD) |
| SPONSOR: | F. Hoffmann-La Roche Ltd. |

## **OBJECTIVES**

## **Primary:**

The primary objective of this study is as follows:

 To evaluate the efficacy of RO6867461 compared to ranibizumab monotherapy in treatment-naive and anti-vascular endothelial growth factor (VEGF)-incompleteresponder patients with CNV secondary to AMD.

## Secondary:

The secondary objectives of this study are as follows:

- To assess the safety of multiple intravitreal (IVT) doses of RO6867461
- To assess systemic pharmacokinetics of RO6867461
- To investigate pharmacodynamics (PD) and anatomical outcomes informing on the mechanism of action of RO6867461
- · To investigate the formation of plasma anti-RO6867461 antibodies
- To investigate 2 different RO6867461 dosing regimens

## **Exploratory:**

The exploratory objectives of this study are as follows:

- To evaluate RO6867461 effects on plasma levels of markers of angiogenesis and inflammation
- To investigate RO6867461 concentration and, if sample volume allows, inflammatory and pro-anglogenic factors, in aqueous humor samples (optional) and vitreous (optional)
- To evaluate the effect of genetic polymorphisms in genes associated with AMD and/or involved in angiogenesis and response to RO6867461

#### STUDY DESIGN

#### **Description of Study**

Multiple-center, multiple-dose and regimen, randomized, active comparator controlled, double-masked, five parallel group, 36-week study in patients with CNV secondary to AMD The five groups of this study are as follows:

- Arm A: 0.5 mg ranibizumab IVT every 4 weeks for 32 weeks (9 injections)
- Arm B: 1.5 mg RO6867461 IVT every 4 weeks for 32 weeks (9 injections)
- Arm C: 6 mg RO6867461 IVT every 4 weeks for 32 weeks (9 injections)
- Arm D: 6 mg RO6867461 IVT every 4 weeks up to Week 12 (4 injections), followed by 6 mg RO6867461 IVT every 8 weeks (i.e., on Weeks 20 and 28; 2 injections)
- Arm E: 0.5 mg ranibizumab IVT every 4 weeks up to Week 8 (3 injections), followed by 6 mg RO6867461 IVT every 4 weeks (6 injections)

The study will allow evaluation of RO6867461 in a treatment-naive patient population (comparison of Arms A, B, C, and D) and an anti-VEGF-incomplete-responder patient population that meets a predefined criterion at Week 12 (comparison between Arms A and E). Only one eye will be chosen as the study eye.

#### **NUMBER OF PATIENTS**

In the initial recruitment period, up to 271 patients with CNV secondary to AMD are expected to be enrolled in the study. Up to 45 (Arms B, C, and D) or 68 (Arms A and E) patients are expected to be randomized per arm of the study (3:2:2:2:3 randomization scheme).

An interim analysis might be conducted to adapt the recruitment up to a maximum of 343 patients in order to have approximately 80 patients in the anti-VEGF-incomplete-responder subgroup completing the study.

#### **TARGET POPULATION**

Male and female patients of ≥50 years of age with treatment-naive CNV secondary to AMD.

#### **INCLUSION/EXCLUSION CRITERIA**

## **Inclusion Criteria:**

Patients must meet the following criteria at study entry:

#### Ocular criteria for study eye:

- Treatment-naïve with CNV secondary to AMD, with subfoveal CNV or juxtafoveal CNV with a subfoveal component related to the CNV activity by fundus fluorescein angiography (FFA) or spectral domain optical coherence tomography (SD-OCT) (such as subretinal fluid, subretinal hyper-reflective material, evidence of leakage, or hemorrhage)
- Best corrected visual acuity (BCVA) letter score of 73 to 24 letters (inclusive) on Early Treatment Diabetic Retinopathy Study (ETDRS)-like charts (20/40 to 20/320 Snellen equivalent) on Day 1. Proportion of patients with BCVA letter score of 73 to 69 letters inclusive (20/40 Snellen equivalent) on Day 1 will be limited to a maximum of 40% of the planned sample size
- CNV lesion of all types (predominantly classic, minimally classic, or occult) with:

Total lesion size (including blood, atrophy, fibrosis, and neovascularization) of  $\leq$ 6 disc areas (DAs) by FFA

CNV component area of ≥ 50% of total lesion size by FFA

Active CNV confirmed by FFA (evidence of leakage)

CNV exudation confirmed by SD-OCT (presence of fluid)

 Clear ocular media and adequate pupillary dilatation to allow acquisition of good quality retinal images to confirm diagnosis

#### General Criteria:

- Able and willing to provide written informed consent and to comply with the study
  protocol according to International Conference on Harmonization (ICH) and local
  regulations. Alternatively, a legally authorized representative must be able to consent
  for the patient according to the ICH and local regulations
- Age ≥50 years
- For women who are not postmenopausal (i.e., ≥ 12 months of non-therapy-induced amenorrhea or surgically sterile (absence of ovaries and/or uterus) agreement to remain abstinent or use combined contraceptive methods that result in a failure rate of <1% per year during the treatment period and at least through Week 36.

Examples of contraceptive methods with an expected failure rate of <1% per year include male sterilization, hormonal implants, proper use of combined oral or injected hormonal contraceptives, and certain intrauterine devices. Alternatively, two methods (e.g., two barrier methods such as a condom and a cervical cap) may be combined to achieve a failure rate of <1% per year, barrier methods must always be supplemented with the use of a spermicide.

- Males must agree to use a barrier method of contraception starting from first treatment administration for at least 2 months post-last treatment administration.
- Patients must be willing not to participate in any other clinical trial including an investigational medicinal product (IMP) or device up to completion of the current study.

#### **Exclusion Criteria:**

Patients who meet any of the following criteria will be excluded from study entry:

#### Ocular criteria for study eve:

- CNV due to causes other than AMD, such as ocular histoplasmosis, trauma, pathological myopia, angioid streaks, choroidal rupture, or uveitis
- Central serous chorioretinopathy (CSC) at screening
- · Retinal pigment epithelial tear involving the macula
- On FFA

Subretinal hemorrhage of >50% of the total lesion area and/or that involves the fovea

Fibrosis or atrophy of >50% of the total lesion area and/or that involves the fovea

- Any prior or concomitant treatment for CNV including (but not restricted to) IVT treatment (steroids, anti-VEGF, transplasminogen activator, ocriplasmin, C<sub>3</sub>F<sub>8</sub> gas, air), periocular pharmacological intervention, argon LASER photocoagulation, verteporfin photodynamic therapy, diode laser, transpupillary thermotherapy, or surgical intervention
- Cataract surgery within 3 months of baseline assessments
- Any other intraocular surgery (pars plana vitrectomy, glaucoma surgery, corneal transplant, radiotherapy)
- Prior IVT treatment (including anti-VEGF medication) except for management of cataract complication with steroid IVT treatment
- Prior periocular pharmacological intervention for other retinal diseases

## Concurrent Ocular Conditions:

- Any concurrent intraocular condition in the study eye (e.g., amblyopia, aphakia, retinal
  detachment, cataract, diabetic retinopathy or maculopathy, or epiretinal membrane with
  traction, etc.) that, in the opinion of the Investigator, could either reduce the potential for
  visual improvement or require medical or surgical intervention
- Active intraocular inflammation (grade trace or above) in the study eye
- · Current vitreous hemorrhage in the study eye
- Uncontrolled glaucoma (e.g., progressive loss of visual fields or defined as intraocular pressure [IOP] ≥25 mmHg despite treatment with anti-glaucoma medication) in the study eye
- Spherical equivalent of refractive error demonstrating more than 8 diopters of myopia in

the study eye

- History of idiopathic or autoimmune-associated uveitis in either eye
- · Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye

#### Characteristics for fellow eye:

- Any anti-VEGF treatment within 7 days prior to Day 1
- Any retinal condition that, in the opinion of the Investigator, might require anti-VEGF treatment within 7 days from Day 1

#### General Criteria:

- Any major illness or major surgical procedure within one month before screening
- Patients with glycosylated hemoglobin HbA1C>7.5%
- Uncontrolled blood pressure ([BP] defined as systolic > 180 mmHg and/or diastolic BP > 100 mmHg while patient at rest). If a patient's initial reading exceeds these values, a second reading may be taken either 30 or more minutes later on the same day, or on another day during the screening period. If the patient's BP is controlled by antihypertensive medication, the patient should be taking the same medication continuously for at least 30 days prior to Day 1
- Stroke within 12 months prior to Day 1
- History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory findings giving reasonable suspicion of a condition that contraindicated the use of the investigational drug or that might affect interpretation of the results of the study or renders the patient at high risk for treatment complications in the opinion of the Investigator
- For females of childbearing potential, a positive blood pregnancy test
- Lactating women
- Known hypersensitivity to ranibizumab, fluorescein, indocyanine green, any ingredients
  of the formulation used, dilating eye drops, or any of the anesthetic and antimicrobial
  drops used
- · Any other restriction accorded to the use of
- Any treatment with an IMP in the 3 months prior to Day 1

## **LENGTH OF STUDY**

The total duration of the study for each patient will be up to 40 weeks, divided as follows:

- Screening: up to 4 weeks
- · Baseline: Day 1
- Study Treatment Administration: from Day 1 to Week 32
- Final safety and efficacy period: from Week 32 to Week 36

#### **END OF STUDY**

The end of the study is defined as the date when the last patient last observation (LPLO) occurs. LPLO is expected to occur 36 weeks after the last patient is enrolled.

#### **OUTCOME MEASURES**

#### SAFETY OUTCOME MEASURES

#### Adverse events

Adverse events and concomitant medications will be monitored throughout the entire study. **Vital signs** 

Body temperature (oral or tympanic) will be collected at the time-points indicated in the schedule of assessments (SoA).

BP and pulse rate will be performed after the patient has rested for at least 5 minutes at the time-points indicated in the SoA.

#### Electrocardiograms

12-lead triplicate electrocardiogram (ECG) will be performed at the time-points indicated in the SoA.

#### Ocular safety

Visual acuity will be assessed using best correction determined from protocol refraction (BCVA) using ETDRS-like charts, slit lamp examination, dilated binocular indirect high-magnification ophthalmoscopy, IOP, fundus photography, SD-OCT, and angiography will be performed at the time-points indicated in the SoA.

#### Laboratory tests

Hematology, blood chemistry, and urinalysis, listed below, will be collected at the time-points indicated in the SoA.

- Hematology: Hemoglobin, hematocrit (HCT), red blood cell count, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), platelet count, total and differential white blood cell count (neutrophils, lymphocytes, monocytes, eosinophils, and basophils in absolute numbers), erythrocyte sedimentation rate (ESR)
- Coagulation (at screening only): Activated partial thromboplastin time (APTT) and prothrombin time/International Normalized Ratio (PT/INR)
- Blood chemistry: Sodium, potassium, bicarbonate, phosphate, chloride, calcium, urea, creatinine, total bilirubin, alkaline phosphatase (ALP), aspartate aminotransferase (AST), alanine aminotransferase (ALT), creatine phosphokinase (CPK), gamma glutamyl transferase (GGT), total protein, glucose, HbA1C (at screening and at final or early termination visits only), total cholesterol (TC), triglycerides (TG), C-reactive protein (CRP)
- Urinalysis: A midstream, clean-catch urine specimen will be collected for dipstick
  analysis of protein, blood, glucose, and pH. Microscopy to be performed if
  abnormalities are observed and deemed necessary by the Investigator or Designee, in
  particular when blood or protein is positive or strong positive
- Pregnancy test: for females of childbearing potential, serum pregnancy test at screening

## Anti-drug antibodies

Plasma samples will be collected at the time-points indicated in the SoA to evaluate the presence of anti-RO6867461 antibodies.

## PHARMACOKINETIC OUTCOME MEASURES

#### Plasma levels of RO6867461

Plasma concentrations will be measured by a specific enzyme-linked immunosorbent assay (ELISA) method. The pharmacokinetic (PK) analysis is described in the statistical methods section. Samples may also be analyzed for ranibizumab.

## Aqueous humor samples (optional)

Samples will be collected from patients who provide additional (optional) consent to participate in aqueous humor collection. Samples will be analyzed for RO6867461 and biomarker concentrations. Samples may also be analyzed for ranibizumab.

## Unscheduled collection of vitreous samples (optional)

If elective vitrectomy surgery is medically necessary, a vitreous sample can be obtained from the study eye from patients who provide additional (optional) consent to participate in vitreous collection for the measurement of RO6867461 and biomarker concentrations.

Samples may also be analyzed for ranibizumab. A blood sample for PK measurement should be taken at the same time.

#### **EFFICACY OUTCOME MEASURES**

The primary efficacy outcome measure for this study is the mean change from baseline BCVA at Week 36 using the ETDRS-modified charts.

The secondary efficacy outcome measures for this study include BCVA and anatomical PD imaging measures relevant to the mechanism of action of RO6867461 as follows:

#### **BCVA**

- Proportion of patients gaining ≥15 letters from baseline BCVA at Week 36
- Proportion of patients with BCVA of 20/40 or better at Week 36
- Proportion of patients with BCVA of 20/200 or worse at Week 36

#### Anatomic outcome measures using SD-OCT

- Mean change from baseline in foveal center point thickness at Week 36
- Mean change from baseline in mean central subfield thickness (1 mm diameter) at Week 36
- Proportion of patients with no intraretinal fluid, subretinal fluid, cysts, or pigment epithelial detachment at Week 36

#### Anatomic outcome measures using FFA

- Mean change from baseline in total area of CNV at Week 36
- · Mean change from baseline in total area of CNV component at Week 36
- Mean change from baseline in total area of leakage at Week 36

#### **EXPLORATORY OUTCOME MEASURES**

The exploratory outcome measures for this study include but are not limited to the following:

- Biomarkers in plasma related to angiogenesis and inflammation
- Pro-angiogenic factors in aqueous humor and vitreous samples for patients who provide consent to participate

## **BIOMARKER/GENOTYPING SAMPLE COLLECTION**

#### **Biomarkers Plasma Samples**

All patients who have been enrolled in the study will have mandatory PD and exploratory biomarker plasma samples taken at the time-points indicated in the SoA. The PD and exploratory plasma samples will be collected to investigate biomarkers in plasma related to angiogenesis and inflammation.

#### Clinical Genotyping (CG) Samples

A mandatory whole blood sample will be taken for DNA extraction from every subject. The DNA may be used to study genes related to AMD (e.g., AMRS2. HTRA1, CFH, C3, etc.) as well as related to angiogenesis (e.g., VEGFA, VEGFR2, angiopoietin-2, angiopoietin-1 receptor [Tie-2], etc.), and the effect on the PK/PD/efficacy/safety of RO6867461. Data arising from this sample will be subject to the same confidentiality as the rest of the study. This specimen will be destroyed no later than 2 years after the final closure of the clinical database.

## **INVESTIGATIONAL MEDICINAL PRODUCT(S)**

IMPs will include the two study drugs as follows:

- RO6867461: Vials of sterile, colorless to brownish, preservative-free solution of RO6867461 (120 mg/mL), for IVT administration of either 1.5 or 6 mg dose every 4 or 8 weeks
  - Placebo is provided as sterile, colorless to slightly brownish, preservative-free liquid, used only for dilution of RO6867461 drug product to the appropriate clinical dose.
- Comparator—Ranibizumab: Vials containing ranibizumab solution (10 mg/mL), for IVT administration of a 0.5 mg dose every 4 weeks.

The double-masked design is achieved through strict independence of the pharmacist (or designated personnel) and Investigators who are preparing and administering study

treatment, from the assessing Investigators and remaining site personnel.

#### NON-INVESTIGATIONAL MEDICINAL PRODUCTS

 Sham: Sham IVT administration will be delivered to patients in Arm D at Weeks 16, 24, and 32 to maintain double-masking throughout the study period.

#### **PROCEDURES**

Detailed SoA and procedures are tabulated in Appendix 1 and Appendix 2 of the protocol.

#### Screening

Treatment-naive patients with CNV secondary to AMD who are willing to participate in the study and have given informed consent will undergo a thorough screening examination within 4 weeks of study treatment administration. The screening procedures as outlined in the SoA will include review of inclusion and exclusion criteria, medical history, physical examination, assessment of vital signs and ECG, serum pregnancy test for female of childbearing potential, and safety laboratory parameters. Imaging criteria for eligibility will be confirmed by a Central Reading Center before enrolment.

#### Treatment period

On Day 1, baseline assessments will be conducted on the eligible patients, according to the SoA. Patients will receive their first IVT administration of either RO6867461 or comparator therapy according to the randomization schedule and following established standard procedures. Patients will return to the eye clinic for study treatment administration (every 4 weeks) and assessments as outlined in the SoA. Patients will be administered the same study treatment throughout the study period, except for the patients randomized to Arms D and E:

- Patients in Arm D will receive sham administrations on Weeks 16, 24, and 32 to maintain the double-masking throughout the every 8 weeks (Q8W) regimen period.
- Patients in Arm E will initially receive 3 injections of ranibizumab followed by 6 injections of RO6867461.

A post-treatment administration check of study eye will be performed for each patient immediately after treatment administration, by testing finger count vision, or hand motion and light perception. On the day of dosing, IOP will be monitored at 30 minutes post-treatment administration in the study eye, and if IOP ≥30 mmHg, IOP should be reassessed at 1 hour post-treatment administration. If IOP continues to be elevated, treatment should be undertaken at the discretion of the Investigator.

#### Final period

Patients will return for final visits with assessments as outlined in the SoA 4 weeks after the last study treatment administration.

## STATISTICAL METHODS

## **SAFETY ANALYSES**

All patients who receive at least one administration of the study treatment will be included in the safety analysis. The safety data, including adverse events, reasons for withdrawal from study, laboratory data, concomitant medications, vital signs, and physical examination results will be listed and summarized descriptively.

As appropriate, listings, summary tables, and graphs (subject plot and/or mean plots) will be provided for safety and tolerability assessments.

Anti-RO6867461 antibody results (positive/negative) will be listed.

General adverse events will be listed and summarized by body system and preferred term using MedDRA. Ophthalmologic adverse events will be listed and summarized.

For laboratory data subject listings will be presented with abnormalities flagged.

#### PHARMACOKINETIC ANALYSES

A nonlinear mixed effects modeling approach (with NONMEM software) will be used to analyze the concentration-time data of RO6867461. Population and individual primary PK parameters (i.e., clearance and volumes) will be estimated and the influence of various covariates (e.g., gender, body weight, etc.) on these parameters will be investigated. The

data collected in this study may be pooled with data collected in the previous Phase I study as appropriate to build a PK model. Secondary PK parameters such as area under the concentration-time curve (AUC) and maximum plasma concentration observed (C<sub>max</sub>) will be derived from the individual post-hoc predictions. The results of this analysis will be reported in a separate document from the clinical study report.

## **PHARMACODYNAMIC ANALYSES**

Individual and mean PD data and parameters will be presented by listings and descriptive summary statistics including means, geometric means, medians, ranges, standard deviations, and coefficients of variation.

An empirical drug-disease model of longitudinal BCVA previously developed on the ranibizumab database will be used to analyze the effect of RO6867461 on BCVA using a meta-analysis approach by integrating data from this study and ranibizumab clinical data.

A similar modeling approach will be used to analyze the relationship between RO6867461 exposure and BCVA. The influence of various baseline covariates on model parameters will be investigated. The PK/PD or dose/PD relationship will be characterized. The results will be reported in a separate document from the clinical study report.

## SAMPLE SIZE JUSTIFICATION

## Sample size and power for treatment-naive population evaluation

The sample size is based on the primary efficacy outcome of BCVA mean change from baseline to Week 36. Each RO6867461 dose or dose regimen group (Arms B, C, and D) will be compared to the control group (Arm A).

The power calculation is based on 68 patients randomized to Arm A, and 45 randomized to each of Arms B, C, and D, with drop-out rate of 10%. Assuming a standard deviation of 13.5 letters, this sample size would provide approximately 80% power to detect a true difference of 5.9 letters at the one-sided  $\alpha$  level of 10%. The minimum detectable difference would be approximately 3.5 letters.

#### Sample size and power for anti-VEGF-incomplete-responder population evaluation

The sample size is based on the primary efficacy outcome of BCVA mean change from Week 12 to Week 36 in the subset of anti-VEGF-incomplete-responders, between Arm A and Arm E.

The power calculation is based on 68 patients randomized to both Arms A and E, with 65% meeting the criteria for inclusion in anti-VEGF–incomplete-responder subgroup and a drop-out rate of 10%. Assuming a standard deviation of 9.7 letters, this sample size would provide around 80% power to detect a true difference of 4.7 letters at the one-sided  $\alpha$  level of 10%. The minimum detectable difference would be approximately 2.7 letters.

#### PRIMARY ENDPOINT ANALYSIS

Evaluation in the treatment naive population: The primary efficacy variable is the mean BCVA change from baseline to Week 36. The primary efficacy analysis will be performed using a Mixed Model for Repeated Measurement (MMRM) model.

Evaluation in the anti-VEGF-incomplete-responder population: The primary efficacy variable is the mean BCVA change from Week 12 to Week 36. The primary efficacy analysis will be performed using a MMRM model.

#### **INTERIM ANALYSES**

An interim analysis may be conducted to allow for adapting the sample size.

An interim analysis of efficacy may be conducted for administrative reasons.

Up to two additional interim analyses may be conducted for efficacy.

## **OTHER CONSIDERATIONS**

N/A

## **LIST OF PROHIBITED MEDICATIONS**

#### Concomitant therapy

Patients who use maintenance therapy other than those required to treat  $wet\ AMD$  (wAMD) should continue its use.

The decision to administer antimicrobial drops before and after the IVT administration is at the discretion of the Investigator.

#### Excluded therapy

At the discretion of the Investigator, patients may continue to receive all medications and standard treatments administered for other conditions except in the following instances:

- · Concurrent use of systemic anti-VEGF agents
- Concurrent use of IVT anti-VEGF therapy in the fellow eye within 7 days before or after study eye treatment
- Concurrent use of IVT or subtenon corticosteroids in either eye, except as required to treat adverse events
- Concurrent use of photocoagulation or photodynamic therapy with verteporfin in the study eye for neovascular AMD

Appendix 2
Schedule of Accessments

| | | | | | Ø | cheduk | of Ass | Schedule of Assessments | ts | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Week | Screening | , M | Week 1 | Week 4 | Week 8 | Week 12 | Week 13 | Week 16 | Week 20 | Week 24 | Week 28 | Week 32 | Week<br>36<br>Final<br>Visit | Early<br>Termination<br>Visit | Unscheduled |
| Day | D-28 to D- | Day<br>1 | Day 7 | Day 28 | Day 56 | Day 84 | Day 91 | Day 112 | Day 140 | Day 168 | Day 196 | Day 224 | Day<br>252 | | |
| Visit Window | | | +-3 | +/-3 | +4-3 | +/-3 | -4/+3 <sup>m</sup> | +/-3 | +/-3 | +-3 | +/-3 | +/-3 | +/-3 | +7 | |
| Assessments | | | | | | | | | | | | | | | |
| Informed Consent | × | | | | | | | | | | | | | | |
| Eligibility | x | Xª | | | | | | | | | | | | | |
| Demography | × | | | | | | | | | | | | | | |
| Medical History | × | × | | | | | | | | | | | | | |
| Physical<br>Examination | × | | | | | | | | | | | | × | × | |
| Anthropometric<br>Measurements | × | | | | | | | | | | | | × | × | |
| Vital Signs | × | 74 | × | 2 | 2 | 2 | × | 2 | 2 | 2 | 2 | 2 | × | × | × |
| ECG-12 lead | × | | | | | | | | | | | | × | × | × |
| Hematology | × | | | | | × | | | | | | | × | × | × |
| Blood Chemistry | × | | | | | × | | | | | | | × | × | × |
| Urinalysis | × | | | : | | × | | | | | | | × | × | × |
| Coagulation | × | | | | | | | | | | | | | | × |
| Pregnancy Test | × | | | | | | | | | | | | | | × |

| Week | Screening | * | Week 1 | Week 4 | Week 8 | Week 12 | Week 13 | Week 16 | Week 20 | Week 24 | Week 28 | Week 32 | Week<br>36<br>Final<br>Visit | Early<br>Termination<br>Visit | Unscheduled |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day | D-28 to D- | Day<br>1 | Day 7 | Day 28 | Day 56 | Day 84 | Day 91 | Day 112 | Day 140 | Day 168 | Day 196 | Day 224 | Day<br>252 | | |
| Visit Window | | | +/-3 | +/-3 | +/-3 | +/-3 | -4/+3 <sup>m</sup> | +/-3 | +1-3 | +1-3 | +4-3 | +4-3 | +/-3 | 2+ | |
| Assessments | X<br>N E | | | | | | | | | | | | | | |
| Administration of Study Medication | | × | | × | × | × | | x<br>or<br>sham | × | x<br>or<br>sham | × | x<br>or<br>sham | | | |
| Safety Finger<br>Count Vision | | × | | × | × | × | | × | × | × | × | × | | | |
| IOP <sup>b, θ</sup> | × | J. K. | × | _<br>(n) | _ლ | ص <sub>ا</sub> | × | ص<br>ا | 3- | 3, | S | 3 | × | × | × |
| BCVA <sup>B,6</sup> | × | × | | × | × | × | | × | × | × | × | × | × | × | × |
| LLVA <sup>®</sup> | | × | | | | × | | | | | | | × | × | × |
| Slit Lamp <sup>a,e</sup> | × | ×ķ | × | × | × | × | × | × | × | × | × | × | × | × | × |
| Ophthalmoscopy | × | × | × | × | × | × | × | × | × | × | × | × | × | × | × |
| Fundus<br>Photography | × | X <sup>k</sup> | | | | × | | | | | : | | × | × | × |
| Fundus<br>Autofluorescence <sup>a</sup> | × | | | i<br>i | | × | | | | | | | × | × | |
| SD-OCT <sup>a</sup> | × | × | × | × | × | × | × | × | × | × | × | × | × | × | × |
| Fundus<br>Fluorescein<br>Angioraphy | × | | | | | × | | | | | | | × | × | × |
| IndoCyanine<br>Green<br>Angiography <sup>a</sup> | × | | | | | × | | | | | | | × | × | |

RO6867461 (VEGF/Ang2)—F. Hoffmann-La Roche Ltd Statistical Analysis Plan BP29647, Version 1

| j | 1 | | 1 | | 1 | | | | | 1 | 1 | 1 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Unscheduled | | | | × | × | | × | × | | × | × | × |
| Early<br>Termination<br>Visit | | +7 | | × | × | | | ! | | × | × | × |
| Week<br>36<br>Final<br>Visit | Day<br>252 | +/-3 | | × | × | × | | | | × | × | × |
| Week 32 | Day 224 | +/-3 | | | | | × | | | | × | × |
| Week 28 | Day 196 | +/-3 | | | | | | | | | × | × |
| Week 24 | Day 168 | +/-3 | 1911 | × | × | × | | | | × | × | × |
| Week 20 | Day 140 | +/-3 | | | | | | | | | × | × |
| Week 16 | Day 112 | +/-3 | | × | × | | | | | × | × | × |
| Week 13 | Day 91 | -4/+3 <sup>m</sup> | | × | × | | | | | | × | × |
| Week 12 | Day 84 | +/-3 | | × | × | × | × | | | × | × | × |
| Week 8 | Day 56 | +/-3 | | | | | | | | | × | × |
| Week 4 | Day 28 | +/-3 | | × | × | × | | | | × | × | × |
| Week 1 | Day 7 | +/-3 | W | | | | | | | | × | × |
| <b>8</b> | Day<br>1 | | | × | × | × | × | | × | × | × | × |
| Screening | D-28 to D-<br>1 | | | | | | | | | | × | × |
| Week | Day | Visit Window | Assessments | PK Sample <sup>a</sup> | PD Biomarkers<br>Sample <sup>a</sup> | Exploratory<br>Plasma Biomarker<br>Sample <sup>a</sup> | Aqueous Humor<br>Sample<br>(optional) <sup>a,d,f,g</sup> | Vitreous Humor +<br>Blood Samples<br>(optional) | Clinical<br>Genotyping<br>Sample <sup>a,i,j</sup> | Anti-Drug<br>Antibody (ADA) <sup>a</sup> | Adverse Events <sup>a</sup> | Previous and Concomitant Treatments |

- Assessment prior to drug administration on days where study treatment is administered
- Multiple assessments on a single visit day, details on timing on a separate table
- Finger count vision assessment asap after, and within maximum of 15 min from study treatment administration
- Assessment in study eye only
- Performed prior to pupil dilation
- Optional sample. Additional consent required from the patient
- Unscheduled sample could be obtained at other or additional planned visits at the discretion of the Investigator in agreement with the participating patient
- Only in case of vitrectomy surgery during the study and if vitreous sampling is feasible. A blood sample for plasma preparation should be drawn at the same time
- Mandatory, except in countries where IRB/EC does not approve.
- At Day 1 but can be done at any other visit if the sample not collected at baseline.
- Baseline assessments
- 1 Assessment post-treatment administration in study eye only
- n Relative to the previous study treatment administration date (Week 12)

# Appendix 3 Definition of ATE

ATE events are non-fatal stroke, non-fatal myocardial infarction, or vascular death (including deaths of unknown cause). They are defined as the following MedDRA terms/baskets:

## Myocardial infarction

SMQ Broad | Myocardial infarction (SMQ)

- PT | Coronary arterial stent insertion
- PT | Coronary artery bypass
- PT | Coronary endarterectomy
- PT | Coronary revascularisation

## Non-myocardial arterial thromboembolic events (ATEs)

- SMQ Narrow | Haemorrhagic cerebrovascular conditions
- SMQ Narrow | Ischaemic cerebrovascular conditions
- PT | Amaurosis
- PT | Amaurosis fugax
- PT | Aortic bypass
- PT | Aortic embolus
- PT | Aortic surgery
- PT | Aortic thrombosis
- PT | Aortogram abnormal
- PT | Arterectomy
- PT | Arterectomy with graft replacement
- PT | Arterial bypass operation
- PT | Arterial graft
- PT | Arterial occlusive disease
- PT | Arterial stent insertion
- PT | Arterial therapeutic procedure
- PT | Arterial thrombosis
- PT | Arteriogram abnormal
- PT | Arteriogram carotid abnormal
- PT | Atherectomy
- PT | Blindness transient
- PT | Carotid angioplasty
- PT | Cerebral hypoperfusion
- PT | Coeliac artery occlusion
- PT | Embolia cutis medicamentosa
- PT | Embolism
- PT | Embolism arterial
- PT | Endarterectomy
- PT | Femoral artery embolism
- PT | Femoral artery occlusion
- PT | Hepatic artery embolism
- PT | Hepatic artery occlusion
- PT | Hepatic artery thrombosis
- PT | Hypothenar hammer syndrome

- PT | Iliac artery embolism
- PT | Iliac artery occlusion
- PT | Intra-aortic balloon placement
- PT | Intraoperative cerebral artery occlusion
- PT | Leriche syndrome
- PT | Mesenteric arteriosclerosis
- PT | Mesenteric artery embolism
- PT | Mesenteric artery stenosis
- PT | Mesenteric artery stent insertion
- PT | Mesenteric artery thrombosis
- PT | Microembolism
- PT | Penile artery occlusion
- PT | Percutaneous coronary intervention
- PT | Peripheral arterial occlusive disease
- PT | Peripheral arterial reocclusion
- PT | Peripheral artery angioplasty
- PT | Peripheral artery bypass
- PT | Peripheral artery stent insertion
- PT | Peripheral artery thrombosis
- PT | Peripheral embolism
- PT | Peripheral endarterectomy
- PT | Popliteal artery entrapment syndrome
- PT | Pulmonary artery therapeutic procedure
- PT | Pulmonary artery thrombosis
- PT | Pulmonary endarterectomy
- PT | Renal artery angioplasty
- PT | Renal artery occlusion
- PT | Renal artery thrombosis
- PT | Renal embolism
- PT | Splenic embolism
- PT | Stress cardiomyopathy
- PT | Subclavian artery embolism
- PT | Subclavian artery occlusion
- PT | Subclavian artery thrombosis
- PT | Superior mesenteric artery syndrome
- PT | Thromboembolectomy
- PT | Thrombotic microangiopathy
- PT | Thrombotic thrombocytopenic purpura
- PT | Truncus coeliacus thrombosis
- PT | Visual acuity reduced transiently

## Venous thromboembolism

- PT | Axillary vein thrombosis
- PT | Budd-Chiari syndrome
- PT | Catheterisation venous
- PT | Cavernous sinus thrombosis
- PT | Central venous catheterisation
- PT | Cerebral venous thrombosis
- PT | Compression stockings application
- PT | Deep vein thrombosis

- PT | Deep vein thrombosis postoperative
- PT | Embolism
- PT | Embolism venous
- PT | Hepatic vein occlusion
- PT | Hepatic vein thrombosis
- PT | Homans' sign positive
- PT | Iliac vein occlusion
- PT | Inferior vena cava syndrome
- PT | Inferior vena caval occlusion
- PT | Intracranial venous sinus thrombosis
- PT | Intravenous catheter management
- PT | Jugular vein thrombosis
- PT | May-Thurner syndrome
- PT | Mesenteric vein thrombosis
- PT | Obstetrical pulmonary embolism
- PT | Obstructive shock
- PT | Ovarian vein thrombosis
- PT | Paget-Schroetter syndrome
- PT | Pelvic venous thrombosis
- PT | Penile vein thrombosis
- PT | Phlebectomy
- PT | Phleboplasty
- PT | Portal vein cavernous transformation
- PT | Portal vein occlusion
- PT | Portal vein thrombosis
- PT | Post procedural pulmonary embolism
- PT | Post thrombotic syndrome
- PT | Postoperative thrombosis
- PT | Postpartum venous thrombosis
- PT | Pulmonary embolism
- PT | Pulmonary infarction
- PT | Pulmonary microemboli
- PT | Pulmonary thrombosis
- PT | Pulmonary vein occlusion
- PT | Pulmonary veno-occlusive disease
- PT | Pulmonary venous thrombosis
- PT | Renal vein embolism
- PT | Renal vein occlusion
- PT | Renal vein thrombosis
- PT | SI QIII TIII pattern
- PT | Splenic vein occlusion
- PT | Splenic vein thrombosis
- PT | Subclavian vein thrombosis
- PT | Superior sagittal sinus thrombosis
- PT | Superior vena cava syndrome
- PT | Thrombophlebitis
- PT | Thrombophlebitis migrans
- PT | Thrombophlebitis neonatal
- PT | Thrombophlebitis superficial
- PT | Thrombosed varicose vein
- PT | Thrombosis corpora cavernosa

- PT | Transverse sinus thrombosis
- PT | Vascular graft
- PT | Vena cava embolism
- PT | Vena cava filter insertion
- PT | Vena cava thrombosis
- PT | Venogram abnormal
- PT | Venoocclusive disease
- PT | Venoocclusive liver disease PT | Venous occlusion
- PT | Venous operation
- PT | Venous recanalisation
- PT | Venous stent insertion
- PT | Venous thrombosis
- PT | Venous thrombosis in pregnancy
- PT | Venous thrombosis limb
- PT | Venous thrombosis neonatal